CLINICAL TRIAL: NCT05750459
Title: Exposure-Response Evaluation of IV Artesunate in Children With Severe Malaria
Brief Title: Pharmacokinetic Study of IV Artesunate to Treat Children With Severe Malaria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-0007; 5UM1AI148689-03 (NIH)
Record Dates: First submitted 2023-02-20; First posted 2023-03-01 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-10-09

CONDITIONS: Plasmodium Falciparum Infection
Keywords: Artesunate; Children; IV; P. falciparum; Severe Malaria; Uganda
MeSH Terms: conditions — Malaria | interventions — Artesunate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Arm 1 (Experimental): Participants will receive the standard of care with IV artesunate for treatment of severe malaria. Each 60-mg vial of artesunic acid will be dissolved in 1 mL of 5% sodium bicarbonate to form sodium artesunate and then mixed with 5 mL of 5% dextrose. This will be injected as a bolus into an indwelling IV cannula. Children weighing <20 kg will receive IV artesunate at a dose of 3.0 mg/kg/dose compared to older children weighing >/= 20kg who will receive 2.4 mg/kg/dose, at times 0, 12, 24. If unable to take oral medication, IV artesunate will continue at 48 and 72 hours. Children who recover and are able to transition to oral antimalarial therapy after a minimum of 24 hours, will initiate a 3-day course of oral artemisinin-combination therapy per national guidelines. N = 100
  Interventions: Drug: Artesunate

INTERVENTIONS:
Drug: Artesunate — Artesunate is a succinic ester of artemether.

SUMMARY:
This clinical study is a phase 4, single-site, open-label pharmacokinetic (PK) study of IV artesunate in up to 100 Ugandan children 6 months-14 years of age who are diagnosed with severe malaria according to standardized World Health Organization (WHO) criteria (any P. falciparum parasitemia and the presence of danger signs). Participants will receive the standard of care IV artesunate for initial treatment of severe malaria per WHO guidelines: children weighing <20 kg should receive 3.0 mg/kg/dose compared to children weighing =20 kg who should receive 2.4 mg/kg/dose, at times 0, 12, 24, 48 and 72 hours (WHO 2015). Parenteral treatment will be administered for a minimum of 24 hours (irrespective of the patient's ability to tolerate oral medication earlier), after which patients will be evaluated clinically and assessed for ability for oral intake of antimalarials. Children who are able to transition to oral antimalarial therapy will initiate a 3-day course of artemisinin-combination oral therapy per national guidelines. The primary objective of the study is to determine the relationship between DHA exposures following IV artesunate dosing and markers of physiologic dysfunction associated with severe malaria in Ugandan children.

DETAILED DESCRIPTION:
This clinical study is a phase 4, single-site, open-label pharmacokinetic (PK) study of IV artesunate in up to 100 Ugandan children 6 months-14 years of age who are diagnosed with severe malaria according to standardized World Health Organization (WHO) criteria (any P. falciparum parasitemia and the presence of danger signs). Participants will receive the standard of care IV artesunate for initial treatment of severe malaria per WHO guidelines: children weighing <20 kg should receive 3.0 mg/kg/dose compared to children weighing =20 kg who should receive 2.4 mg/kg/dose, at times 0, 12, 24, 48 and 72 hours (WHO 2015). Parenteral treatment will be administered for a minimum of 24 hours (irrespective of the patient's ability to tolerate oral medication earlier), after which patients will be evaluated clinically and assessed for ability for oral intake of antimalarials. Children who are able to transition to oral antimalarial therapy will initiate a 3-day course of artemisinin-combination oral therapy per national guidelines. Biomarkers of physiologic dysfunction will be quantified at regular intervals, including serum lactate, serum glucose, total and direct bilirubin, bicarbonate levels, Blantyre Coma Score (BCS), creatinine and hemoglobin. These biomarkers will be considered both independently and together as a weighted score to relate to the PK of the active metabolite of IV artesunate, DHA and to efficacy markers that more accurately reflect clinical outcomes. We will also quantify P. falciparum parasitemia using standardized thick blood smear and relate this outcome to DHA dose and exposure for comparison with historical studies. Children 6 months to 14 years of age living in or near Tororo District, Uganda, who are diagnosed with severe malaria and who meet inclusion and exclusion criteria will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Children ages 6 months-14 years at the time of severe malaria diagnosis, inclusive
2. Meet the case definition for severe malaria, per WHO standardized guidelines
3. Parent/guardian willing to provide informed consent
4. Assent for children between 8 and 14 years who are conscious and otherwise able to provide assent, inclusive

Exclusion Criteria:

1. Receipt of > 24 hours of artemisinin therapy

Ages: 6 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline bicarbonate levels | Day 1 through Day 183
Change from baseline creatinine. | Day 1 through Day 183
Change from baseline diastolic blood pressure | Day 1 through Day 183
Change from baseline in Blantyre Coma Score (BCS). | Day 1 through Day 183
Change from baseline in concentration of Dihydroartemisinin (DHA) | Day 1
  Pharmacokinetic parameters that will be derived from the concentration of Dihydroartemisinin (DHA) include maximum concentration (C max), area under the curve over hours 0-12 (AUC 0-12) and half-life (t 1/2) and time to C max (T max).
Change from baseline in direct bilirubin | Day 1 through Day 183
Change from baseline in hemoglobin | Day 1 through Day 183
Change from baseline in serum glucose | Day 1 through Day 183
Change from baseline in temperature. | Day 1 through Day 183
Change from baseline in total bilirubin | Day 1 through Day 183
Change from baseline in venous serum lactate. | Day 1 through Day 183
Change from baseline systolic blood pressure | Day 1 through Day 183

SECONDARY OUTCOMES:
Parasite (P. falciparum) density in thick blood smear. | Day 1 through Day 5 minimum
  Parasite clearance as calculated from parasite density over time, as measured by thick blood smear such as parasite clearance half-life, total parasite clearance by Day 2, and time to 90% reduction in parasitemia.
Time to hospital discharge. | Day 1 through 183

CONTACTS AND LOCATIONS:
Locations (1):
- Makerere University-Infectious Diseases Institute, Kampala, Uganda

DOCUMENTS (3):
  • Study Protocol (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT05750459/Prot_001.pdf
  • Statistical Analysis Plan (2025-02-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT05750459/SAP_002.pdf
  • Informed Consent Form (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT05750459/ICF_000.pdf